CLINICAL TRIAL: NCT06509763
Title: ElectrocardioGraphic Imaging During Left bUndle Branch Implant to valiDate Ecg Criteria
Acronym: GUIDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, Arrhythmia Section MD PhD, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GUIDE
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: Electrocardiographic Imaging; Left Bundle Branch Pacing; Cardiac Resynchronization Therapy; Conduction System Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Left Bundle Branch electrode implant (Experimental)
  Interventions: Device: ECGI system during LBBP implant

INTERVENTIONS:
Device: ECGI system during LBBP implant — ECGI system to create non-invasive ventricular maps during the screwing steps of the LBBP electrode

SUMMARY:
The goal is to validate the resynchronization criteria with a non-invasive technique, during the LBBP implant. Non-invasive real-time ventricular activation maps will be created and analyzed before, during, and after the implantation of the left bundle branch lead, including right septal pacing, mid and deep septal pacing and pacing when reaching the left bundle branch according to the published standard LBBP criteria. Using these maps, the investigators will quantify activation times and evaluate changes in the ventricular sequence during implantation.

ELIGIBILITY:
Inclusion Criteria:

* Left bundle branch pacing indication
* Capability of standing up to place the ECGI vest

Exclusion Criteria:

* Less than 18 years-old
* Patients with cognitive impairment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Left ventricular resynchronization assessed by ECGI | During procedure
  Resynchronization assesed by non-invasive ECGI by the Left Ventricle Activation Time reduction and the septal activation ventricular pattern once reaching the LBBP according to the published ECG criteria.

SECONDARY OUTCOMES:
VEU | During procedure
  Ventricular Electrical Uncoupling computed as the difference between the mean activation time of the left and the right ventricle
LVDI | During procedure
  Left Ventricle Dyssinchrony Index computed as the standard deviation of individual activations recorded from the left ventricle.
Histogram Overlap | During procedure
  Overlapping of the right ventricle and left ventricle activation times histogram distributions as a parameter to assess the dyssinchrony between ventricles.
LVAT | During procedure
  Left Ventricular Activation Time computed as the difference between the earliest and the latest actvation of the left ventricle
Isochronal Crowding | During procedure
  Number of Isochrones presented in the left ventricular activation map to assess the homogeneity of the activation

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Tolosana, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona; Margarida Pujol, MD, PhD, Study Director — Hospital Clinic of Barcelona; Lluis Mont Girbau, MD,PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang W, Huang J, Qi Y, Wang F, Guo L, Shi X, Wu W, Zhou X, Li R. Cardiac resynchronization therapy by left bundle branch area pacing in patients with heart failure and left bundle branch block. Heart Rhythm. 2019 Dec;16(12):1783-1790. doi: 10.1016/j.hrthm.2019.09.006. Epub 2019 Sep 9. PMID 31513945
- [Background] Cai B, Huang X, Li L, Guo J, Chen S, Meng F, Wang H, Lin B, Su M. Evaluation of cardiac synchrony in left bundle branch pacing: Insights from echocardiographic research. J Cardiovasc Electrophysiol. 2020 Feb;31(2):560-569. doi: 10.1111/jce.14342. Epub 2020 Jan 20. PMID 31919928
- [Background] Zhang S, Zhou X, Gold MR. Left Bundle Branch Pacing: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Dec 17;74(24):3039-3049. doi: 10.1016/j.jacc.2019.10.039. Epub 2019 Dec 9. PMID 31865972
- [Background] Wu S, Chen X, Wang S, Xu L, Xiao F, Huang Z, Zheng R, Jiang L, Vijayaraman P, Sharma PS, Su L, Huang W. Evaluation of the Criteria to Distinguish Left Bundle Branch Pacing From Left Ventricular Septal Pacing. JACC Clin Electrophysiol. 2021 Sep;7(9):1166-1177. doi: 10.1016/j.jacep.2021.02.018. Epub 2021 Apr 28. PMID 33933414
- [Background] Huang W, Chen X, Su L, Wu S, Xia X, Vijayaraman P. A beginner's guide to permanent left bundle branch pacing. Heart Rhythm. 2019 Dec;16(12):1791-1796. doi: 10.1016/j.hrthm.2019.06.016. Epub 2019 Jun 22. No abstract available. PMID 31233818
- [Background] Ploux S, Lumens J, Whinnett Z, Montaudon M, Strom M, Ramanathan C, Derval N, Zemmoura A, Denis A, De Guillebon M, Shah A, Hocini M, Jais P, Ritter P, Haissaguerre M, Wilkoff BL, Bordachar P. Noninvasive electrocardiographic mapping to improve patient selection for cardiac resynchronization therapy: beyond QRS duration and left bundle branch block morphology. J Am Coll Cardiol. 2013 Jun 18;61(24):2435-2443. doi: 10.1016/j.jacc.2013.01.093. Epub 2013 Apr 16. PMID 23602768
- [Background] Elliott MK, Blauer J, Mehta VS, Sidhu BS, Gould J, Jackson T, Sieniewicz B, Niederer S, Ghosh S, Rinaldi CA. Comparison of electrical dyssynchrony parameters between electrocardiographic imaging and a simulated ECG belt. J Electrocardiol. 2021 Sep-Oct;68:117-123. doi: 10.1016/j.jelectrocard.2021.08.003. Epub 2021 Aug 8. PMID 34416669